CLINICAL TRIAL: NCT03095170
Title: Physical Exercise And Cognitive Engagement Outcomes for Mild Neurocognitive Disorder
Acronym: PEACEOFMND
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB Closure
Sponsor: University of Florida (Other)
Collaborators: Mayo Clinic (Other); Tallahassee Memorial HealthCare (Other); Florida Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201700004; 7AZA1 (Other Grant/Funding Number: Florida Department of Health); 9AZ15 (Other Grant/Funding Number: Florida Department of Health); IRB201900522 (Other: UF (PEACEOFMND Extension)); OCR21041 (Other: UF OnCore)
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Mild Cognitive Impairment; Memory Disorders; Mild Dementia; Impaired Cognition; Mild Cognitive Disorder; Amnestic Disorder; Dementia and Amnestic Conditions; Poor Short-term Memory; Memory Impairment; Mild Neurocognitive Disorder
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders; Cognition Disorders; Neurocognitive Disorders; Dementia | interventions — Yoga; Self-Help Groups; Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Computerized brain fitness training (Experimental): Will receive a 10 day intervention program (over 2 weeks) consisting of Computer Brain Fitness Training, Calendar Training and Support Group.
  After the initial two week intervention, there will be an extended period during which participants will continue the computerized brain fitness for another 24 weeks.Participants are encouraged to do at least two hours per week.
  Interventions: Behavioral: Computerized brain fitness training; Behavioral: Support Group (patient and partner); Behavioral: Cognitive Rehabilitation
- Yoga (Experimental): Will receive a 10 day intervention program (over 2 weeks) consisting of Yoga, Calendar Training, and Support Group.
  After the initial two week intervention, there will be an extended period during which participants will continue yoga for 24 weeks. Participants assigned to the yoga intervention will continue to meet with their group and their yoga instructor for one hour per week and will be expected to do at least an additional hour of yoga by themselves every week.
  Interventions: Behavioral: Yoga; Behavioral: Support Group (patient and partner); Behavioral: Cognitive Rehabilitation
- Wellness Education (Active Comparator): Will receive a 10 day intervention program (over 2 weeks) consisting of Wellness Education, Calendar Training and Support Group.
  Interventions: Behavioral: Wellness Education; Behavioral: Support Group (patient and partner); Behavioral: Cognitive Rehabilitation

INTERVENTIONS:
Behavioral: Computerized brain fitness training — Will use the commercially available Posit Science product BrainHQ™ (www.brainhq.com) on tablets (e.g. iPads). Participants will complete 45-60 minutes of training daily in the program.
  Other Names: Brain Fitness
  Arms: Computerized brain fitness training
Behavioral: Yoga — Will use adapted Hatha Yoga where participants sit on armless chairs placed on sticky mats for some asana (poses) and use the chair for support throughout. This adapted Hatha Yoga style is appropriate for older adults including those who have limited mobility, use walkers or are in wheelchairs. The appropriately sequenced yoga practice meets the American College of Sports Medicine recommendation for older adults for muscle strengthening and flexibility. Instructions are modeled for the participants
  Arms: Yoga
Behavioral: Wellness Education — The education component will involve daily 60-minute group sessions with topics such as Introduction to the Program, Living with MCI, Changes in Roles, Communication and Relationships, Sleep Hygiene, Steps to Healthy Brain Aging, Preventing Dementia, MCI and Depression, Nutrition, Safety and Assistive Technologies, and Participating in Research, Community Resources, Meaning and Purpose, and Joy.
  Arms: Wellness Education
Behavioral: Support Group (patient and partner) — Journal© as a basis for reminiscence-focused group sessions. Partner: The care partner support group meets separately from the patient group for 45-60 minutes daily.
Behavioral: Cognitive Rehabilitation — Will provide each couple with memory compensation training 5 days per week for 2 weeks, with initial and ending adherence sessions. All sessions will involve 45- 60 minutes of training. The curriculum is described briefly here.
  Learning phases. three training stages from learning theory: 1) an acquisition phase in which use of the memory compensation system is learned, 2) an application phase in which a participant is taught to apply to his/her daily life, and 3) an adaptation phase in which a participant practices incorporating into his/her daily life so as to make its use habitual.
  Other Names: Memory Compensation Training; Memory Support System

SUMMARY:
Behavioral interventions currently provide the most useful approach to addressing the behavioral and social needs of those with Mild Cognitive Impairment (MCI) due to Alzheimer's or other diseases. This randomized, multisite, 3-arm study will investigate the impact of computerized brain fitness vs yoga vs an active control group (wellness education) on changes in cognitive function, daily functioning and quality of life in persons with Mild Cognitive Impairment (MCI) and their partner. In addition, in vivo neuroimaging measures of plasticity during the pre- and post-intervention periods will be measured and compared between the three different treatment groups. These neuroimaging measures of plasticity will be investigated in their relationship to the cognitive outcomes within each group.

ELIGIBILITY:
For the patients diagnosed with MCI:

Inclusion Criteria:

1. Written informed consent for participation. Patient also needs to sign a legally authorized representative (LAR) addendum should MCI patient become incapacitated
2. A diagnosis of amnestic MCI (single domain or multi-domain)
3. A Clinical Dementia Rating scale score of 0 or 0.5
4. At least 50.
5. Either not taking or stable on nootropic(s) and/or pain medication for at least 3 months.
6. Fluent in English.
7. A score of at least 25 on the Telephone Interview for Cognitive Status for Memory.

Exclusion Criteria:

1. MRI contraindications (e.g., ferrous metal in the body, claustrophobia, pregnancy)
2. Physical impairments, language comprehension deficits, or significant hearing disturbances that would limit ability to perform tasks or participation in the intervention.

For the care partners:

Inclusion Criteria:

1. Written informed consent for participation.
2. At least 21 years of age.
3. A score of at least 32 on the Telephone Interview for Cognitive Status for Memory.
4. Partner has at least twice-weekly contact with the participant.

Exclusion Criteria:

1. Physical impairments, language comprehension deficits, or significant hearing disturbances that would limit ability to perform tasks or participation in the intervention.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Resting State Magnetic Resonance Imaging (MRI) | baseline to 7.5 months
  Resting State MRI will allow us to investigate the functional connectivity in the brain, by looking at resting state networks such as the Default Mode Network.

SECONDARY OUTCOMES:
Diffusion Tensor Imaging (DTI) | baseline to 7.5 Months
  DTI will be used to map white matter tractography in the brain.

OTHER OUTCOMES:
improvement in patient memory based everyday functioning | baseline to 7.5 Months
  measured by the Everyday Cognitive Functioning scale (ECOG)
improvement in patient and care partner quality of life | baseline to 7.5 Months
  measured by the quality of life measured by the Quality of Life in Alzheimer's Disease scale (QOL-AD)
improvement in patient and carepartner mood | baseline to 7.5 Months
  measured by the Center for Epidemiological Studies-Depression (CESD)
improvement in patient cognitive functioning | baseline to 7.5 Months
  measured by the CogState

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Smith, Ph. D, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Wit L, O'Shea D, Chandler M, Bhaskar T, Tanner J, Vemuri P, Crook J, Morris M, Smith G. Physical exercise and cognitive engagement outcomes for mild neurocognitive disorder: a group-randomized pilot trial. Trials. 2018 Oct 19;19(1):573. doi: 10.1186/s13063-018-2865-3. PMID 30340619